CLINICAL TRIAL: NCT06606431
Title: Accompaniment of Isolated People by Volunteers From the Neighborhood: a Community Mixed Quasi-experimental/Qualitative Clinical Trial
Brief Title: ACOMPANYEM: A COMmunity Program Accessing Lonely, Disabled Neighbors (Young, Elder, and Midlife)
Acronym: ACOMPANYEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Sara Martínez Torres, Research Technician, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24/095-P (Ethics Committee nº)
Record Dates: First submitted 2024-09-05; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Social Isolation or Loneliness; Homebound Persons; Disabled Persons
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Pre-Post Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Group (Experimental): The intervention is multilevel and is based on bringing together two population groups in the community with complementary needs:
  1. People over 16 years of age isolated at home due to mobility problems or chronic mental illness.
  2. Volunteers from the neighborhood, especially people with interested in improving their emotional well-being.
  REBEC will conduct a first individual interview to confirm that the volunteers are emotionally and vitally stable at the time of the intervention.
  A personalized relational dynamic of help will be set up in each case (one-to-one interaction, relational level). This interaction can consist of listening at home or going with the person on the street to bring them closer to the different proposals for community social activities.
  The group of social isolation and/or unwanted loneliness will also receive support from the community team, to provide a personalized response to the physical, health, social or psychological needs detected by the v
  Interventions: Behavioral: Multileveled-community approach
- Control Group (No Intervention): In-waiting list for intervention in future rounds; habitual care

INTERVENTIONS:
Behavioral: Multileveled-community approach — One-to-one delivered interaction at relational level (Interpersonal Relations, Volunteers) Socio-health interaction at personalized level (Social Work) Group delivered interaction for volunteers (Group Dynamics) Community-level interactions (Social Cohesion, Community Networks)
  Arms: Participant Group

SUMMARY:
Social prescription prioritizes interventions for people at risk of social isolation or unwanted loneliness based on community assets and offers them a series of activities that can contribute to their emotional well-being as a healthy alternative to medicalized healthcare. Disabled homebound people deal with more difficulty accessing the social health assets available in the community. Volunteers from the same neighborhood may accomplish the social function of accompaniment and listening accessing them at home or walking them out to attain social prescription goals. The Community Emotional Well-Being Referent (REBEC) may enhance all of this by conducting emotional counseling and management groups for volunteers.

OBJECTIVE: To evaluate the effectiveness of a community intervention of accompaniment and emotional management with volunteers on the unwanted loneliness of people with social isolation, their emotional well-being, and their quality of life.

METHODOLOGY: a community-based quasi-experimental non-randomized pre-post intervention study with control group, and a qualitative study. Candidate detection by the Driving Group, composed of neighborhood organizations and the community health team, was conducted opportunistically. Recruitment of isolated individuals and volunteers was carried out, with registration based on inclusion criteria. Implementation of the multi-level intervention for volunteers and isolated individuals took place at home or by participating in community resources on the street, with parallel support groups for volunteers using REBEC. Each round of participants was followed for three months, continuing until the sample was complete. Qualitative analysis was conducted upon reaching information saturation. In cases where architectural barriers were detected, technical aids (such as portable stairlifts) were proposed, and their impact was studied.

ELIGIBILITY:
Inclusion Criteria:

Previously detected by community and professional assets among people over 16 years of age with the following criteria:

* Disabled physical or mental homebound persons.
* Unwanted loneliness, with difficulty in accessing other assets of the social prescription program.
* less than 8 on the Oslo Social Support Scale or less than 20 on the LSNS-R scale or less than 2 on the LSNR-6 scale in people over 65 years of age.

Exclusion Criteria:

* Impossibility of communication
* End-of-life situations.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Social Support/Isolation | 3 months for each round
  Social Support Scale (OSLO 3) (Kocalevent, 2018).
  The Oslo 3 social support scale is part of the ECHI list (European Community Health Indicators). Study the relationship between support and psychological suffering. It consists of three questions:
  * How many people do you have around when you need them because you have a severe problem? Outcomes: 0, 1-2, 3-5, 5+.
  * What interest do people show in what you do? Answers: many, some, uncertain, little, not at all.
  * Is it easy for you to ask your neighbors for help if you need it? Answers: quite easy, easy, possible, difficult, exceedingly difficult.
  The result of the scale is the sum of the score of all the questions. The range is between 3 and 14 points. Outcome classifies as follows:
  * Between 3 and 8: poor social support.
  * Between 9 and 11: medium social support.
  * Between 12 and 14 high social support.
Emotional Well-Being | 3 months for each round
  Emotional Well-being Scale (7 items) SWEMWBS (Castellví, 2017). The questionnaire consists of seven items measured with a Likert-type scale, with five answer options (1 never - 5 always), about how the person has felt in the last two weeks. This questionnaire has recently been adapted to Catalan and Spanish and added to the Catalan Health Survey.
  The result of the emotional well-being test is the sum of the score of each item. Therefore, the score ranges from 5 to 35.
  There are no cut-off points. Well-being is a continuum, and we cannot consider itself high, medium, or low. The interesting thing is to see the evolution of well-being in the same person.
Loneliness | 3 months
  Unwanted loneliness will be addressed separately in a qualitative study as a complex and empirical phenomenon, not guided from the outset by predetermined theories (constructivist perspective). It will be measured in a semi-structured interview with a single binary answer question: "Do you feel lonely?" (yes/no). This will be followed by a Visual Analogue Scale to attempt to measure the subjective feeling of loneliness, which could be more associated with poor psychological health than with the perception of a reduction in the number of relationships. Additionally, a single question will be used to evaluate whether the person wishes to be accompanied (yes/no), followed by another VAS to measure the extent of this desire.
Health-Related Quality of Life (HRQoL) | 3 months for each round
  The EQ-5D is a HRQoL instrument used both in general population and in groups of patients with diverse conditions. The individual himself assesses his or her state of health, first with descriptive system that values severity of symptoms and then in visual analogue scale (VAS). Ther are five dimensions of health (mobility, personal care, daily activities, pain/discomfort, and anxiety/depression) and each of them has three levels of severity (no problems, problems or moderate problems and serious problems). In this part of the questionnaire, the individual must mark the level of severity corresponding to their state of health in each of the dimensions, referring to the same day that they complete the questionnaire. In each dimension of the EQ-5D, the severity levels are encoded with a 1 if the answer option is (no (have) problems); with a 2 if the answer option is (some or moderate problems); and with a 3 if the answer option is (many problems).
Social Support/Isolation for aged more than 65 | 3 months for each round
  The Lubben Social Network Scale (LSNS) assesses perceived social support and risk of isolation in older adults. Developed by J. Lubben and team, it evaluates the size, proximity, and frequency of social contacts through a brief series of questions, typically taking 10-15 minutes. The LSNS-R has 12 items, split between family and non-family contacts, and provides four results: three subscales for perceived social support (family, non-family, global; ranges 0-30, 0-60) and one for risk of isolation. Scores reveal risk levels: low (more than 30), moderate (26-30), high (21-25), and social isolation (less than 20). The LSNS-6, a shorter version with six items, covers family and non-family relations and yields two results: perceived social support (range 0-30) and risk of isolation (score ≤12) (Lubben et al., 2006; Pérez Pavilla, 2021)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Atenció Primària Bonavista-La Canonja. Gerència Territorial Camp de Tarragona, Institut Català de la Salut, Barcelona, Spain, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No